CLINICAL TRIAL: NCT02694016
Title: Remote Ischemic Preconditioning in Patients Undergoing Isolated Aortic Valve Replacement Surgery With a Biological Prosthesis: A Single Center Randomized Prospective Study
Brief Title: Remote Ischemic Preconditioning in Patients Undergoing Isolated Aortic Valve Replacement Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment pace
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Fredrik Yannopoulos, Resident, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RIPC00AVR
Record Dates: First submitted 2016-02-18; First posted 2016-02-29 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Aortic Valve Disease; Myocardial Ischemia
Keywords: Remote ischemic preconditioning; Neuroprotection
MeSH Terms: conditions — Aortic Valve Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Experimental): Patient will undergo normal isolated aortic valve replacement surgery with a biological prosthesis and a preoperative lower leg remote ischemic preconditioning(RIPC) phase.
  Interventions: Procedure: Remote ischemic preconditioning
- Control group (No Intervention): Patient will undergo normal isolated aortic valve replacement surgery with a biological prosthesis

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — A blood pressure cuff is placed around the right leg on the level of the thigh. Randomization is performed after this, using sealed envelopes with covariate balancing for age and sex. Regardless of the outcome of the randomization the cuff is left in place so as not to give any indication of which group the patient belongs to. If the patient is randomized into the remote ischemic preconditioning group (RIPC) then four (4) cycles of five (5) minute inflation are given after induction. Each cycle is followed by a five (5) minute interval of reperfusion. Cuff pressure should be 200mgHg at least (RRsyt + 100mmgHg) during the inflation periods.
  Arms: Remote ischemic preconditioning

SUMMARY:
The goal is to investigate the efficacy, safety and possible neuro- and cardioprotective effects of remote ischemic preconditioning (RIPC) in adult cardiac patients undergoing isolated aortic valve replacement surgery with a biological prosthesis. Neuropsychological evaluation preoperatively and at 30d after surgery will establish if there are any differences in neuropsychological performance between groups. A large array of biochemical markers will be analyzed from plasma samples taken at different time points. Additionally skin biopsies from the lower limb will be taken before and after performing RIPC on said limb. During the venous cannulation phase a atrial biopsy will be taken. The biochemical markers from plasma and tissue samples will be used to asses brain tissue damage, inflammation and cardiac tissue damage between groups.

This will be a single center prospective randomized study with two groups. A intervention group (RIPC) and a control group. Study size is: 40 patients in total, 20 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Non-emergency aortic valve replacement with a biological prosthesis with perfusion and cardiac arrest

Exclusion Criteria:

* Recent myocardial infarction
* Carotid stenosis requiring intervention
* Any other concomitant surgical procedure
* Increased troponin baseline before surgery
* Critical ischemia of lower limbs
* Peripheral arterial disease (ASO, media sclerosis)
* Morbid obesity (Incompatible cuff-to-thigh diameter)
* Severe heart insufficiency
* Moderate to severe venous insufficiency lower limbs
* Recent acute stroke <90d
* Difference in cardioplegic protocol
* Diseased aorta in epiaortic ultrasound

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Neuropsychological assesment | 1 month postoperatively
  Investigators will use a neuropsychological test battery to test our subject pre- and post-operatively. A qualified psychologist will administer the test battery. The test battery will be relatively simple but still have several different tests. These tests will include but are not limited to:
  - Trail Making test A & B (TMT)
Neuropsychological assesment | 1 month postoperatively
  Digit Span test
Neuropsychological assesment | 1 month postoperatively
  Rey Auditory Verbal Learning Test (RAVLT)

SECONDARY OUTCOMES:
Inflammation markers analysed from plasma and tissue samples | A day before surgery, during surgery, 24hour and 48hour postoperatively
  A bioplex/multiplex assay of systemic inflammatory response markers and other cytokines including but not limited to:
  Tumor Necrosis Factor-a, Interleukin-1b, -2, -4, -5, -6. C-Reactive Protein, Hypoxia inducible Factor -1.
Tissue specific markers analysed from plasma | A day before surgery, during surgery, 24hour and 48hour postoperatively
  A bioplex/multiplex assay of neuronal and cardiac tissue specific biomarkers including but not limited to:
  S-100b, Glial Fibrillary acidic protein, Neuron Specific enolase, Troponin-I, Brain Natriuretic Peptide, Creatinine Kinase - MB

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Yannopoulos, MD Ph.D, Study Director — Oulu University Hospital; Vesa Anttila, MD Ph.D., Study Chair — Oulu University Hospital; Tuomas Ahvenvaara, MD, Principal Investigator — Oulu University Hospital; Tuomas Mäkelä, MD.Ph.D., Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Department of Cardiothoracic surgery, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No